CLINICAL TRIAL: NCT05507372
Title: Treatment for Post Acute COVID-19 Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Applied Biology, Inc. (Industry)
Collaborators: Jupiter Wellness, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JW-COVID-DRG-001
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus | interventions — Pimozide

STUDY DESIGN:
Intervention Model Description: Blinded, placebo controlled parallel assignment randomised study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dopamine Receptor Modulator (Experimental): Pimozide 1mg Oral
  Interventions: Drug: Pimozide 1 MG
- Placebo (Placebo Comparator): Placebo Oral
  Interventions: Drug: Pimozide 1 MG

INTERVENTIONS:
Drug: Pimozide 1 MG — Dopamine Receptor Antagonist - Oral Pimozide

SUMMARY:
Post-acute COVID-19 tinnitus has not been treated successfully. As tinnitus may be related to SARS-CoV-2 neurological manifestations. This study aims to investigate if the dopamine receptor antagonists can be used effectively treat COVID-19 induced tinnitus.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is the causative viral pathogen leading to the COVID-19 pandemic. In 2022, after three successive waves of the pandemic, the majority of the human population has been exposed to the SARS-CoV-2 virus. During the two years since the pandemic ensued, multiple reports emerged of patients experiencing COVID-19 emergent symptoms lasting longer than 4 weeks since onset. Up to 15% of patients recovering from COVID-19 experience post-acute COVID-19 induced tinnitus .

To-date, post-acute COVID-19 tinnitus has not been treated successfully. As tinnitus may be related to SARS-CoV-2 neurological manifestations. This study aims to investigate if the dopamine receptor antagonist Pimozide can be used effectively treat COVID-19 induced tinnitus.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with subjective tinnitus post COVID-19
2. Tinnitus persists for at least 4 weeks
3. Prior history of mild or no tinnitus
4. 18 years or older
5. Any gender
6. Females of child bearing age must be on contraception

Exclusion Criteria:

1. Pregnant
2. Patients who participated in any interventional studies in the past 6 months
3. Patients with severe hepatic impairment on admission (alanine aminotransferase higher than fivefold the upper limit)
4. Patients taking any dopamine receptor antagonists
5. Patient having history of hypersensitivity to Pimozide
6. Patients unable to comply with the study schedule
7. Actively using cortiocosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | 4 weeks
  The Tinnitus Handicap Inventory Scale is between 0-100. And is stratified to Grades between 1-5. A higher grades means more severe handicap from tinnitus.

CONTACTS AND LOCATIONS:
Overall Officials: RAHUL RAJENDRA KUNKULOL, MBBS, Principal Investigator — DEPT.OF PHARMACOLOGY, RURAL MEDICAL COLLEGE, PIMS- DU (DU), LONI, PIN: 413736

IPD SHARING:
Plan to Share IPD: No